CLINICAL TRIAL: NCT06547021
Title: Investigating the Effect of Different Frequencies of Transcranial Electrical Stimulations Paired With Cognitive Training on the Executive Brain Functions in Dementia Population
Brief Title: Investigating Different Frequencies of Transcranial Electrical Stimulations in Dementia Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HS26590 (B2024:091)
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-08

CONDITIONS: Dementia
Keywords: transcranial electrical stimulation
MeSH Terms: conditions — Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: All participants receive all 4 treatments in a randomized order with washout period of 2-5 months. After finishing all 4 treatments, participants receive one more treatment protocol after the washout period where the participant will receive tACS at the personalized gamma over the regular placement of electrodes (left dorsolateral prefrontal cortex and the reference electrode on the contralateral supraorbital area) for the first 30-min training session and then over the precuneus (one electrode over Pz on the 10-20 EEG system and the other over the right deltoid muscle) during the second 30-min training session. Once they complete the Pz protocol, participants will receive their optimal treatment with the first 30-min targeting the left DLPFC and the second 30-min targeting the right DLPFC (one electrode over right DLPFC and one over contralateral supraorbital area).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The order of treatments is only known by the study coordinator, the PI and the supervisor. The order of treatments will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- Transcranial Direct Current Stimulation (tDCS) (Experimental): Participants will receive tDCS simultaneously with cognitive exercises for one month every day excluding weekends.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Gamma Transcranial Alternating Current Stimulation (tACS) (Experimental): Participants will receive personalized gamma tACS simultaneously with cognitive exercises for one month every day excluding weekends.
  Interventions: Device: Gamma Transcranial Alternating Current Stimulation (tACS)
- Theta Transcranial Alternating Current Stimulation (tACS) (Experimental): Participants will receive personalized theta tACS simultaneously with cognitive exercises for one month every day excluding weekends.
  Interventions: Device: Theta Transcranial Alternating Current Stimulation (tACS)
- Sham Stimulation (Experimental): Participants will receive sham stimulation simultaneously with cognitive exercises for one month every day excluding weekends.
  Interventions: Device: Sham
- Gamma Transcranial Alternating Current Stimulation (tACS)-Precuneus (Experimental): Participant will receive tACS at the personalized gamma over the regular placement of electrodes (left dorsolateral prefrontal cortex and the reference electrode on the contralateral supraorbital area) for the first 30-min training session and then over the precuneus (one electrode over Pz on the 10-20 EEG system and the other over the right deltoid muscle) during the second 30-min training session.
  Interventions: Device: Gamma Transcranial Alternating Current Stimulation (tACS)-Precuneus
- Bilateral DLPFC (Experimental): Applying the optimal tES over left and right DLPFC. First 30-min will target the left DLPFC similar to the other arms, and the second 30-min treatment will target tES to the right DLPFC (one electrode over right DLPFC and one electrode over contralateral supraorbital area).
  Interventions: Device: Bilateral DLPFC

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — A light electrical current with zero frequency (tDCS) will be applied to the participants' scalp via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. Cognitive exercises will be performed through the "Mind Triggers" app on an iPad where the participants perform memory and learning games/tasks.
  Arms: Transcranial Direct Current Stimulation (tDCS)
Device: Gamma Transcranial Alternating Current Stimulation (tACS) — A light electrical current with personalized gamma frequency (tACS) will be applied to the participants' scalp via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. Cognitive exercises will be performed through the "Mind Triggers" app on an iPad where the participants perform memory and learning games/tasks.
  Arms: Gamma Transcranial Alternating Current Stimulation (tACS)
Device: Theta Transcranial Alternating Current Stimulation (tACS) — A light electrical current with personalized theta frequency (tACS) will be applied to the participants' scalp via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. Cognitive exercises will be performed through the "Mind Triggers" app on an iPad where the participants perform memory and learning games/tasks.
  Arms: Theta Transcranial Alternating Current Stimulation (tACS)
Device: Sham — Sham stimulation (i.e. only slight stimulation at the beginning and at the end for a few seconds with majority of the time having no stimulation) will be applied to the participants' scalp via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. Cognitive exercises will be performed through the "Mind Triggers" app on an iPad where the participants perform memory and learning games/tasks.
  Arms: Sham Stimulation
Device: Gamma Transcranial Alternating Current Stimulation (tACS)-Precuneus — A light electrical current with personalized gamma frequency (tACS) will be applied to the participants' scalp via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. Cognitive exercises will be performed through the "Mind Triggers" app on an iPad where the participants perform memory and learning games/tasks.
  Arms: Gamma Transcranial Alternating Current Stimulation (tACS)-Precuneus
Device: Bilateral DLPFC — A light electrical current applied to the participants' scalp via 2 electrodes, while the participants perform cognitive exercises with the guidance of a trained research assistant. First 30-min treatment will target left DLPFC and second 30-min treatment will target right DLPFC. Cognitive exercises will be performed through the "Mind Triggers" app on an iPad where the participants perform memory and learning games/tasks.
  Arms: Bilateral DLPFC

SUMMARY:
Dementia is a prevalent condition with no known cure. It affects not only the person with dementia but also the family. This study will investigate the effects of applying different transcranial electrical stimulation (tES) waveforms to find the optimal stimulation when paired with cognitive exercise on older adults with dementia. It is a placebo-controlled double-blind study with statistical rigor. In addition, the investigators will investigate technological methods to monitor changes due to the intervention. These include functional near infrared spectroscopy (fNIRS), electroencephalography (EEG), electrovestibulography (EVestG), and balance measurements using accelerometers. fNIRS measures oxygenated and deoxygenated blood flow to the brain and it may help to understand neuronal changes due to intervention. EEG measures the electrical activity of the brain via electrodes placed on the scalp to study the brain's response to different electrical stimulations treatments. EVestG is a non-invasive measure of the vestibuloacoustic system in both background (no motion) and in response to passive whole-body tilt stimuli. We hypothesize there is a direct link between vestibular system deficiencies and Alzheimer's. Lastly, the investigators will measure the effects of electrical stimulation on balance by measuring postural sway using two accelerometers.

This study investigates the effects of transcranial alternating current stimulation (tACS) and transcranial direct current stimulation (tDCS) with different protocols for frequencies to determine the most effective treatment to improve cognitive abilities and working memory for people with dementia.

The global objective of the proposed study is to investigate the effects of different tES in improving the cognitive status of older adults with dementia, when paired simultaneously with cognitive training. The general objectives include the following:

1. Run a human research randomized and double-blind study to address the global objective of the study with statistical rigor.
2. Investigate the correlation of fNIRS outcomes with those of the primary outcome measures of the study in Objective 1 as well as its predictivity to the treatment at baseline.
3. Investigate the effects of different tES on EEG recordings as well as its predictivity to the treatment at baseline.
4. Investigate the effects of different tES on balance for older adults with cognitive impairment.
5. Investigate the correlation of EVestG outcomes with those of the primary outcome measures of the study in Objective 1 as well as its predictively to the treatment at baseline.
6. Disseminate the project results and design the next follow up project.

DETAILED DESCRIPTION:
About 100 participants with either mild cognitive impairment (MCI) or a probable early or moderate dementia type excluding Parkinsonian dementia (as confirmed by their treating physician), will be recruited and tested over the course of this study.

Participants will have the option to choose to do the stimulation and cognitive exercise from home or at Riverview Health Centre. However, all assessments will be completed at Riverview Health Centre. One of the main limitations of human research is the small sample size as recruitment and enrollment of eligible participants especially in dementia population is a major challenge. Thus, a longitudinal study. Each participant will receive all 4 tES protocols in a randomized order while playing cognitive exercises:

1. Personalized gamma tACS
2. Personalized theta tACS
3. tDCS (zero frequency)
4. Sham tES The protocol for all tES treatments will be 4 weeks, 5 days/week (excluding weekends), two 30-min training sessions/day with 15 to 30 min break in between, all tutored either in-person or virtually. Participants will be assessed the week before each new treatment block, within a week of post-treatment and a month after the end of treatment block (follow-up). Between the different tES treatment protocols, 8-week to 20-week washout period will take place with no treatment. The time period for each participant to receive all 4 protocols will be around one year and a half depending on the duration of the washout period. After the participant completes all 4 protocols, there is one more treatment protocol where the participant will receive tACS at the personalized gamma over the regular placement of electrodes (left dorsolateral prefrontal cortex and the reference electrode on the contralateral supraorbital area) for the first 30-min training session and then over the precuneus (one electrode over Pz on the 10-20 EEG system and the other over the right deltoid muscle) during the second 30-min training session. Then the investigators will offer the treatment type (any of the above 5 experimental types) with the highest efficacy for each participant. In other words, the investigators will offer an optimized treatment after the one year and a half.

The eligibility criteria for enrolling individuals into this study are: 50 y<age<95 y, 5<MoCA<24.

Exclusion criteria are any of the followings:

* Being diagnosed with Parkinson's, Parkinsonian dementia, Huntington disease, speech significant aphasia and intellectual disability, major depression/anxiety, bipolar disorder, schizophrenia or any other major mood disorder.
* Having a History of epileptic seizures or epilepsy
* Inability to adequately communicate in English
* Impaired vision or hearing severe enough to impair performance in cognitive tests
* Current substance abuse disorder
* Currently participating in another therapeutic study for dementia

The global objective of the proposed study is to investigate the effects of different tES in improving the cognitive status of older adults with dementia, when paired simultaneously with cognitive training. The general objectives include the following:

1. Run a human research randomized and double-blind study to address the global objective of the study with statistical rigor.
2. Investigate the correlation of fNIRS outcomes with those of the primary outcome measures of the study in Objective 1 as well as its predictivity to the treatment at baseline.
3. Investigate the effects of different tES on EEG recordings as well as its predictivity to the treatment at baseline.
4. Investigate the effects of different tES on balance for older adults with cognitive impairment.
5. Investigate the correlation of EVestG outcomes with those of the primary outcome measures of the study in Objective 1 as well as its predictively to the treatment at baseline.
6. Disseminate the project results and design the next follow up project.

ELIGIBILITY:
Inclusion Criteria:

* MoCA score between 5 and 24
* Between the age of 50 and 95 years old

Exclusion Criteria:

* Being diagnosed with Parkinson's, Parkinsonian dementia, Huntington disease, speech significant aphasia and intellectual disability, major depression/anxiety, bipolar disorder, schizophrenia or any other major mood disorder.
* Having a History of epileptic seizures or epilepsy
* Inability to adequately communicate in English
* Impaired vision or hearing severe enough to impair performance in cognitive tests
* Current substance abuse disorder
* Currently participating in another therapeutic study for dementia
* Change to medication for Alzheimer's disease, dementia, or depression

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale (ADAS-Cog) | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  11 tasks include the participant completing tests and observer based assessments. It assesses cognitive domains of memory, language and praxis. The score ranges from 0 to 70 where higher score indicates greater cognitive impairment.
Wechsler Memory Scale (WMS-IV) | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  Cognitive and memory task that focuses on 6 major memory indexes: auditory memory, visual working memory, immediate memory, delayed memory, and recognition memory. The score ranges from 40 to 160 where the lower score indicates greater cognitive impairment.

SECONDARY OUTCOMES:
Neuropsychiatric Inventory Questionnaire (NPI-Q) | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  Questionnaire used to assess neuropsychiatric symptoms and caregiver burden. The score is based on the presence of a specified symptom and a separate score for severity of the symptom. For presence the minimum total score is 0, maximum score is 12. For severity the minimum total score is 0, maximum is 36. Higher scores indicate participant is exhibiting more severe changes in behaviours.
Montgomery-Asberg Depression Rating Scale (MADRS) | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  Questionnaire which measures mental health and more specifically depression severity where participant rates answers from zero to 6 for 10 questions. The score ranges from 0 to 60 with higher score indicating increased severity of depression.
Functional Near Infrared Spectroscopy (fNIRS) | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  Device designed mainly to measure blood flow over the prefrontal cortex. Participants will perform math and N-back task while fNIRS measures the signals simultaneously.
EEG power in theta band | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9), and pre- and post-treatment EEG for 3 treatments days
  The theta band power will be calculated from each EEG recording.
EEG power in gamma band | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  The gamma band power will be calculated as the average from the tasks performed during EEG recording.
Peak gamma frequency from EEG | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  The peak gamma frequency will be calculated from each EEG recording.
Peak theta frequency from EEG | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  The peak theta frequency will be calculated as the average from the tasks performed during EEG recording.
Postural Sway from balance assessment | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  Postural sway (i.e. peak frequency of sway) will be measured using accelerometers placed on the back and ankle of the participant.
Vestibular Disorders Activities of Daily Living Scale (VADL) | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  VADL (vestibular disorders activities of daily living scale) will be recorded which is a questionnaire with 28 items rated from 1 to 10. Minimum score of 28 with maximum score of 280. This will be used in the analysis of balance data.
BMI | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  Height and weight will be recorded for each participant in order to calculate BMI. This will be taken into account for analyzing balance data.
Width of EVestG signal | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  The width of the action potential from the EVestG signal will be analyzed for changes due changes in vestibular system and its functioning.
Blood Pressure | For each treatment: baseline (week 0), post-treatment (week 5), 1-month follow-up (week 9)
  Blood pressure measurement will be recorded for each participant 3 times. This will be taken into account for analyzing EVestG and fNIRS.

CONTACTS AND LOCATIONS:
Locations (1):
- Riverview Health Centre, Winnipeg, Canada